CLINICAL TRIAL: NCT06602648
Title: Novel Health Care Strategies for Melanoma in Children, Adolescents, and Young Adults. Histological, Computational, and Molecular Pathology for Improved Diagnosis. (Mol-Mel). Work Package 3 (WP3)
Brief Title: MELCAYA - Novel Health Care Strategies for Melanoma in Children, Adolescents, and Young Adults - Work Package 3 (WP3)
Acronym: Mol-Mel
Status: Recruiting | Type: Observational
Sponsor: University of Florence (Other)
Collaborators: Tubingen University Hospital (Unknown); Maria Sklodowska-Curie National Research Institute of Oncology (Other); Fondazione IRCCS ISTITUTO NAZIONALE TUMORI (Unknown); Hospital Clinic of Barcelona (Other); Istanbul University (Other); University Of Perugia (Other); German Cancer Research Center (Other)
Responsible Party: Principal Investigator, Daniela Massi, Professor, University of Florence
Other Study IDs: 24680_bio
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Melanoma of Skin
Keywords: Melanoma; Pediatric; Childrens; Adolescents; Young adults
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Formalin fixed and paraffin embedded (FFPE) samples of melanoma collected from the patient during routine surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CAYA Melanoma patients: Patients under 30 years of age at the moment of melanoma diagnosis. The patients have been divided in Children (1-14 yrs), Adolescents (15-18 yrs) and Young Adults (18-30 yrs) based on the age of diagnosis.

SUMMARY:
The aim of this study is to investigate a type of skin cancer, also known as melanoma, in children, adolescents, and young adults, who will be referred to as CAYA patients in this project. The need for this study arises because this disease, in CAYA patients, is still poorly understood due to its rarity in individuals under 30 years old. This often leads to difficulties in assessing its severity and, consequently, in deciding on the necessary treatments to ensure the patient's recovery. The goal of this study is to examine melanoma in CAYA patients in order to gather the information needed to provide better diagnoses for affected patients and, as a result, select appropriate treatments to fight the disease and promote the patient's full recovery. Additionally, the data collected will be used to create a Pan-European online platform that will allow doctors across the European Union to consult the obtained data and collaborate on particularly complex melanoma cases, always with the aim of ensuring the patient's full recovery in the shortest possible time.

DETAILED DESCRIPTION:
The Mol-Mel study will focus on different tasks and for each task different investigations will be carried out:

* Standardization and tissue quality control: The quality of the samples will then be determined using hematoxylin & eosin (HE)-staining. If any quality issue is detected feedback will be sent to the clinical center responsible for providing the sample
* Histopathology & computational pathology: Melanoma samples will undergo a central pathology review and analysis of conventional prognostic staging parameters. Diagnostically challenging neoplasms will be included in an "inter-observer agreement" carried out by different pathologist.Melanoma samples will also be charactered by single and multi-plex IHC in whole sections and tissue microarrays (TMA), and subjected to automated digital quantification. Spatial proteomics by automated ultra-high content imaging/MACSima Imaging Cyclic Staining (MICS) technology enables simultaneous analysis of hundreds of marker antigens on a single sample. Hundreds of antigens for single sample will be analysed via "Automated ultra-high content imaging/MACSima Imaging Cyclic Staining" (MICS) that will be performed on the novel automated ultra-high content imaging platform MACSimaTM (Miltenyi Biotec).
* Comprehensive somatic, transcriptional and DNA methylation landscape and data integration: DNA and RNA will be extracted by FFPE melanoma samples and characterized using whole-exome sequencing (WES), single nucleotide polymorphism (SNP) and RNA sequencing (RNAseq) arrays on matched tumor/normal pairs of samples. Then recurrent somatic aberrations, DNA methylation subclasses and patterns of tumor evolution will be characterized.
* Pan-European digital second opinion platform: this last task will focus on creating a pan-european second opinion platofrom in order to facilitate standardization of melanoma diagnosis and to share knowledge about biomarkers, algorithms and subtype classification.

ELIGIBILITY:
Inclusion Criteria:

* adolescent and childhood patients (< 20 years) or young adults (< 30 years)
* histologically confirmed diagnosis of melanoma or intermediate/ambiguous melanocytic neoplasm (i.e., melanocytomas, SAMPUS, IAMPUS and MELTUMP according to WHO classification)

Exclusion criteria:

* adult patients (> 30 years of age)
* patients without histologically confirmed diagnosis of melanoma or intermediate/ambiguous melanocytic neoplasm

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will focus on CAYA (< 30 y.o) patients with histologically confirmed melanoma or intermediate/ambiguous melanocytic neoplasm (i.e.,melanocytomas, SAMPUS, IAMPUS and MELTUMP according to WHO classification).The population include patients of both genders.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Primary objective - Hybrid taxonomy | From enrollment at the end of 32 months
  Integrate histopathology and molecular analyses to provide a novel hybrid taxonomy of melanoma in CAYA.
Primay objective - Histopathological and molecular features of pediatric melanoma | From enrollment at the end of 32 months
  Assess the histopathological and molecular features of pediatric melanomas.

SECONDARY OUTCOMES:
Secondary Objective - Identification of biomarkers | From enrollment at the end of 32 months
  Identify prognostic biomarkers in the context of immunotherapy and targeted therapy.
Secondary Objective - pan-European digital pathology platform | From enrollment at the end of 32 months
  Create a pan-European digital pathology platform to assess diagnostic inter-observer reproducibility, enhance international collaboration and achieve diagnosis standardization.
Secondary Objective - Identification of prognostic and predictive biomarkers | From enrollment at the end of 32 months
  Identify driver mutations, transcriptomes, and DNA methylation subclasses with morphological, immunophenotypic analyses and clinical data to provide a novel hybrid taxonomy and identify tissue prognostic and predictive biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Massi Daniela, Principal Investigator — University of Florence (UNIFI)
Locations (1):
- University of Florence, Florence, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Informations about the patients will be shared with other collaborators for the sharing of histological and clinical data in order to reach a consensus diagnosis between collaborating pathologists. Each collected sample will receive a identification code which will allow the results of the automated process to be saved and compared with those noted by the pathological anatomy medical staff. The code is assigned through pseudonymisation techniques (reversible de-identification), so that it cannot be directly traced back to the interested parties.
Supporting Information: ICF
Time Frame: Up to 32 months from enrollment
Access Criteria: The data will be managed by the main investigator of the study: Prof Daniela Massi, according to the recent European regulations in force of the GDPR and the Provision containing the requirements relating to the processing of particular categories of data, pursuant to art. 21, paragraph 1 of Legislative Decree 10 August 2018, n. 101 (GU no. 176 of 29 July 2019).
  Other collaborators can only access histopathological and clinical data of the patients.

REFERENCES:
- [Background] Pappo AS. Melanoma in children and adolescents. Eur J Cancer. 2003 Dec;39(18):2651-61. doi: 10.1016/j.ejca.2003.06.001. PMID 14642927
- [Background] Wiesner T, Kutzner H, Cerroni L, Mihm MC Jr, Busam KJ, Murali R. Genomic aberrations in spitzoid melanocytic tumours and their implications for diagnosis, prognosis and therapy. Pathology. 2016 Feb;48(2):113-31. doi: 10.1016/j.pathol.2015.12.007. Epub 2016 Jan 18. PMID 27020384
- [Background] Barnhill RL, Argenyi ZB, From L, Glass LF, Maize JC, Mihm MC Jr, Rabkin MS, Ronan SG, White WL, Piepkorn M. Atypical Spitz nevi/tumors: lack of consensus for diagnosis, discrimination from melanoma, and prediction of outcome. Hum Pathol. 1999 May;30(5):513-20. doi: 10.1016/s0046-8177(99)90193-4. PMID 10333219
- [Background] Cordoro KM, Gupta D, Frieden IJ, McCalmont T, Kashani-Sabet M. Pediatric melanoma: results of a large cohort study and proposal for modified ABCD detection criteria for children. J Am Acad Dermatol. 2013 Jun;68(6):913-25. doi: 10.1016/j.jaad.2012.12.953. Epub 2013 Feb 8. PMID 23395590
- [Background] de Vries M, Vonkeman WG, van Ginkel RJ, Hoekstra HJ. Morbidity after inguinal sentinel lymph node biopsy and completion lymph node dissection in patients with cutaneous melanoma. Eur J Surg Oncol. 2006 Sep;32(7):785-9. doi: 10.1016/j.ejso.2006.05.003. Epub 2006 Jun 27. PMID 16806794
- [Background] Ferrari A, Brecht IB, Gatta G, Schneider DT, Orbach D, Cecchetto G, Godzinski J, Reguerre Y, Bien E, Stachowicz-Stencel T, Ost M, Magni C, Kearns P, Vassal G, Massimino M, Biondi A, Bisogno G, Trama A. Defining and listing very rare cancers of paediatric age: consensus of the Joint Action on Rare Cancers in cooperation with the European Cooperative Study Group for Pediatric Rare Tumors. Eur J Cancer. 2019 Mar;110:120-126. doi: 10.1016/j.ejca.2018.12.031. Epub 2019 Feb 19. PMID 30785015
- [Background] Saiyed FK, Hamilton EC, Austin MT. Pediatric melanoma: incidence, treatment, and prognosis. Pediatric Health Med Ther. 2017 Apr 18;8:39-45. doi: 10.2147/PHMT.S115534. eCollection 2017. PMID 29388632
- [Background] Jen M, Murphy M, Grant-Kels JM. Childhood melanoma. Clin Dermatol. 2009 Nov-Dec;27(6):529-36. doi: 10.1016/j.clindermatol.2008.09.011. PMID 19880040
- See also: MELCAYA official website — https://www.melcaya.eu/